CLINICAL TRIAL: NCT02837731
Title: Evaluation of Fluid Volume in Patients With Sepsis and Refractory Hypotension
Brief Title: Fluid Responsiveness Evaluation in Sepsis-associated Hypotension
Acronym: FRESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheetah Medical Inc. (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-OOO1
Record Dates: First submitted 2016-07-14; First posted 2016-07-20 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Hypotension
MeSH Terms: conditions — Sepsis; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Starling SV monitor (Experimental): A dynamic assessment of fluid responsiveness using the Starling SV monitor will be performed at every clinical decision point for the first 72 hours of study enrollment. Examples of a clinical decision point include a mean arterial pressure (MAP) of < 65, the decision to give additional fluid volume, and the decision to either escalate or wean vasopressors. Fluid responsiveness will be assessed using a passive leg raise (PLR) to guide corresponding treatment.
  Interventions: Device: Treatment Starling SV monitor
- Control (No Intervention): No required therapeutic protocol will be used for patient treatment, and is determined per the discretion of the physician and hospital standards.

INTERVENTIONS:
Device: Treatment Starling SV monitor — A dynamic assessment of fluid responsiveness will be performed at every clinical decision point for the first 72 hours of study enrollment. Fluid responsiveness will be assessed using a passive leg raise (PLR) and Starling SV hemodynamic monitor to guide corresponding treatment.
  Arms: Treatment Starling SV monitor

SUMMARY:
This study assesses the mean difference in fluid balance at ICU discharge and associated patient outcomes, based on a dynamic assessment of fluid responsiveness in septic patients with refractory hypotension in an ICU setting.

DETAILED DESCRIPTION:
Multi-center randomized study comparing dynamic assessment of fluid responsiveness utilizing Starling SV monitor compared to a control group.

Subjects will be randomized in a 2:1 treatment to control group ratio to increase power for sub-analysis by patient population.

Patients randomized to the Starling SV arm will have treatment guided by a dynamic assessment of fluid responsiveness (measured by a change in stroke volume index > 10%) as assessed by passive leg raise (PLR).

Patients randomized to the control group will receive standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sepsis, as exhibited by 2 or more of the following systemic inflammatory response syndrome (SIRS) criteria and a known or presumed infection at time of screening:

   * Temperature of > 38 C or < 36 C
   * Heart rate of > 90/min
   * Respiratory rate of > 20/min or PaCO2 < 32 mm Hg (4.3 kPA)
   * White blood cell count > 12000/mm3 or < 4000/mm3 or >10% immature bands
2. Refractory hypotension despite initial fluid resuscitation (1L of treatment fluid)
3. Patient enrolled in study as soon as possible (ideal window of 0-12 hours) and within 24 hours of arrival to the hospital
4. Anticipated ICU admission
5. Able to provide signed informed consent or consent can be obtained from the patient's authorized representative

Exclusion Criteria:

1. Primary diagnosis of: acute cerebral vascular event, acute coronary syndrome, acute pulmonary edema, status asthmaticus, major cardiac arrhythmia, drug overdose, or injury from burn or trauma
2. Known aortic insufficiency, or aortic abnormalities
3. Hemodynamic instability due to active gastrointestinal hemorrhage
4. Patient has received >3 liters of IV fluid prior to study randomization
5. Requires immediate surgery
6. Patient transferred to the ICU from another hospital unit
7. Do not attempt resuscitation (DNAR or DNR) order
8. Advanced directives restricting implementation of the resuscitation protocol
9. Contraindication to blood transfusion
10. Attending clinician deems aggressive resuscitation unsuitable
11. Transferred from another in-hospital setting
12. Not able to commence treatment protocol within 1 hour after randomization
13. Known intraventricular heart defect, such as ventral septal defect or atrial septal defect
14. Use of additional hemodynamic monitoring involving stroke volume variation (SVV) to determine fluid responsiveness
15. Seizure in the last 24 hours
16. Prisoner
17. Pregnancy
18. Age <18
19. Known allergy to sensor material or gel
20. Inability or contraindication to doing a passive leg raise with both extremities, such as inability to interrupt venous compression boots
21. Patient has an epidural catheter in place
22. Suspected intra-abdominal hypertension
23. Inability to obtain IV access
24. Diabetic ketoacidosis
25. Hyper-osmolarity syndrome
26. Patient uncouples from treatment algorithm
27. Patient should be excluded based on the opinion of the Clinician/Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (11):
  - University of California San Francisco Medical Center, San Francisco, California
  - Denver Health, Denver, Colorado
  - Grady Memorial Hospital, Atlanta, Georgia
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - NYU School of Medicine, New York, New York
  - New York Presbyterian Brooklyn Methodist Hospital, New York, New York
  - Ohio State University Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Royal Surrey County Hospital, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Summary data will be reviewed periodically

REFERENCES:
- [Derived] Douglas IS, Alapat PM, Corl KA, Exline MC, Forni LG, Holder AL, Kaufman DA, Khan A, Levy MM, Martin GS, Sahatjian JA, Seeley E, Self WH, Weingarten JA, Williams M, Hansell DM. Fluid Response Evaluation in Sepsis Hypotension and Shock: A Randomized Clinical Trial. Chest. 2020 Oct;158(4):1431-1445. doi: 10.1016/j.chest.2020.04.025. Epub 2020 Apr 27. PMID 32353418

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Starling SV Monitor; Usual Care: During Allocation phase, randomization was a 2:1 allocation of SV-guided to usual care. Subjects that didn't complete Follow-up phase are those that (1) show data that indicates unacceptable bias in the measurements, (2) data collection is interrupted prior to 72 hour data collection period of ICU stay, or (3) severe agitation and/or cardiopulmonary resuscitations resulted in poor quality data. Subjects completed follow-up were included in the Analysis.
Period: Allocation
Arm/Group | Treatment Starling SV Monitor | Usual Care
Started | 102 | 48
Completed | 83 | 41
Not Completed | 19 | 7
Not completed — Admitted to General Floor | 3 | 4
Not completed — Immediate surgery/withdrew | 2 | 0
Not completed — Diabetic Ketoacidosis/withdrew | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Device not available | 1 | 0
Not completed — Protocol not implemented | 7 | 0
Not completed — Moribund/Do not resuscitate | 2 | 0
Not completed — Did not meet sepsis criteria | 1 | 2
Not completed — Known aortic abnormalities | 0 | 1
Period: Follow-up
Arm/Group | Treatment Starling SV Monitor | Usual Care
Started | 83 | 41
Completed | 83 | 41
Not Completed | 0 | 0
Period: Analysis
Arm/Group | Treatment Starling SV Monitor | Usual Care
Started | 83 | 41
Completed | 83 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat
Groups:
- Treatment Starling SV Monitor: A dynamic assessment of fluid responsiveness using the Starling SV monitor will be performed at every clinical decision point for the first 72 hours of study enrollment. Examples of a clinical decision point include a mean arterial pressure (MAP) of < 65, the decision to give additional fluid volume, and the decision to either escalate or wean vasopressors. Fluid responsiveness will be assessed using a passive leg raise (PLR) and Starling SV hemodynamic monitor to guide corresponding treatment.
- Usual Care: No required therapeutic protocol will be used for patient treatment, and is determined per the discretion of the physician and hospital standards.
- Total: Total of all reporting groups
Arm/Group | Treatment Starling SV Monitor | Usual Care | Total
Number analyzed (Participants) | 83 | 41 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (16.9) | 62.7 (15) | 62.1 (16.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 13 | 64
  Male | 32 | 28 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 31 | 92
  Black or African American | 17 | 9 | 26
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 1 | 0 | 1
  Unknown | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fluid Balance
Description: Fluid balance is defined as all intravenous fluids administered over a 72 hour period (or ICU discharge, whichever occurred first), minus all fluid output. Urine output was measured in the ICU in 12 hour increments.
Time Frame: 72 hours
Population: mITT population was predefined as including all patients who signed consent, met study eligibility criteria, were randomized and received monitoring for 72 hours or ICU discharge if earlier. mITT (n=83,41).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
Liters | 0.65 (2.85) | 2.02 (3.44)
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Superiority; p = 0.021, t-test, 2 sided; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-2.53 to 0.21]

2. Secondary Outcome: Percentage of Participants Requiring Renal Replacement Therapy
Description: Renal replacement therapy (RRT) is therapy that replaces the normal blood-filtering function of the kidneys. It is used when the kidneys are not working well, which is called kidney failure and includes acute kidney injury and chronic kidney disease. Patient receives new treatment with dialysis.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 79 | 40
percentage of participants | 5.1 | 17.5
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; p = 0.042, Fisher Exact; Mean Difference (Final Values) = -0.124, 95% CI 2-sided [-0.27 to -0.01] — Converted Estimated Value of -12.4% to decimal value of -0.124

3. Secondary Outcome: Percentage of Participants Requiring Ventilator Use
Description: Patients did not enter the study on ventilation, but required ventilator use during the study are included in the analysis.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 79 | 41
percentage of participants | 17.7 | 34.1
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; p = 0.044, Chi-squared; Mean Difference (Final Values) = -0.1642, 95% CI 2-sided [-0.33 to 0] — Converted Estimated Value of -16.42% to decimal value of -0.1642

4. Secondary Outcome: Length of ICU Stay
Description: Intensive Car Unit (ICU) length of stay will be calculated using the earliest of date that the subject is medically ready for discharge when captured, the date of discharge, or the study exit date.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 74 | 35
days | 3.31 (3.51) | 6.22 (10.72)
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; p = 0.113, Fisher Exact; Mean Difference (Final Values) = -2.91, 95% CI 2-sided [-6.67 to 0.85]

5. Secondary Outcome: Number of Hours of Ventilator Use
Description: Patients that did not enter the study on ventilation, but required ventilator use during the study are included in the analysis.Ventilator use might have improved (less use of ventilator support), had no change, or worsened (more use of ventilator support).
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 14 | 14
hours | 46.99 (52.33) | 119.42 (134.90)
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -72.43, 95% CI 2-sided [-154.08 to 9.22]

6. Secondary Outcome: Number of Hours of Vasopressor Use
Description: Vasopressor drugs are provided to restore and maintain blood pressure in patients with septic shock. Patients that have vasopressors initiated throughout the trial are included in this analysis.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 55 | 26
hours | 40.74 (51.23) | 55.64 (87.42)
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; p = 0.426, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -14.91, 95% CI 2-sided [-52.50 to 22.68]

7. Secondary Outcome: Change From Baseline in Serum Creatinine Levels at 72 Hours
Description: The diagnosis of Acute Kidney Injury (AKI) is traditionally based on a rise in serum creatinine
Time Frame: Baseline, 72 hours
Population: mITT
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 79 | 34
mg/dL | 0.13 (1.10) | 0.04 (0.97)
Statistical Analysis 1: Comparison: Treatment Starling SV Monitor vs Usual Care; Test type: Other; p = 0.453, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.34 to 0.52]

8. Other Pre Specified Outcome: Volume of Fluid
Description: Traditional methods of assessing fluid responsiveness (FR) such as vital signs, physical examination, and static measurements of circulatory pressure have shown not to reliably correlate with fluid responsiveness. In contrast, dynamic measurement of stroke volume (SV) following an intravenous (IV) fluid bolus or passive leg raise (PLR) is a safe and feasible method of rapidly assessing the effectiveness of fluid-induced augmentation of SV and cardiac output (CO). Mean volume of treatment fluid Administered (ml) at 72 hours or ICU discharge, whichever occurs first, between the two treatment groups
Time Frame: 72 hours
Population: mITT
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
ml | 5759.2 (2246.8) | 6865.5 (3348.5)

9. Other Pre Specified Outcome: Percentage of Participants With Major Adverse Cardiac Event (MACE)
Description: Incidence of cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
percentage of participants | 6 | 12.2

10. Other Pre Specified Outcome: Number of Participants Experiencing an Adverse Event (AE) Related to Study Device
Description: Adverse events associated with the treatment procedure.
Time Frame: Day 1 to Day 30
Population: ITT-all randomized.
Measure: Number; unit: participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 102 | 48
participants | 1 | 0

11. Other Pre Specified Outcome: Percentage of Participants With Hospital Discharge Without ICU Readmission
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
percentage of participants | 94.9 | 97.8

12. Other Pre Specified Outcome: Percentage of Participants Within Overall 30 Day Mortality Rate
Description: Incidence of death.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
percentage of participants | 15.7 | 22

13. Other Pre Specified Outcome: Number of Participants by Hospital Discharge Location
Description: Patient location (either "home" or "other") following hospital discharge.
Time Frame: Day 1 to Day 30
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Starling SV Monitor | Usual Care
Number analyzed (Participants) | 83 | 41
Participants
  Home | 53 | 18
  Other | 30 | 23

ADVERSE EVENTS:
Time Frame: Day 1 to Day 30
Description: It was not pre-specified in the Study Protocol to collect Other (Not Including Serious) Adverse Events. For Mortality and SAE, safety analyses were performed on randomized (ITT) population.
Arm/Group | Treatment Starling SV Monitor | Usual Care
All-Cause Mortality (participants affected / at risk) | 20/102 | 10/48
Serious Adverse Events (participants affected / at risk) | 10/102 | 7/48
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Starling SV Monitor (N=102) | Usual Care (N=48)
Cardiac Arrest (Cardiac disorders) | 3 (3) | 3 (3)
Intubation/respiratory distress (Cardiac disorders) | 1 (1) | 0 (0)
Severe septic shock and transition to comfort care (Cardiac disorders) | 1 (1) | 0 (0)
Intubation and ards (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intubation and surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress requiring intubation and transfer to ICU (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Multiorgan Failure (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Skin tear and possible infection related to the monitor leads (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Specifics of the publication policy will be outlined to the Investigator in the Clinical Trial Research Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02837731/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02837731/SAP_001.pdf